CLINICAL TRIAL: NCT04768023
Title: Influence of 12 Weeks Vitamin D Supplementation Combined With Physical Activity on Blood and Functional Parameters and Quality of Life in Parkinson's Disease Patients Treated With Deep Brain Stimulation
Brief Title: 12 Weeks Vitamin D Supplementation and Physical Activity in PD Patients With DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: PD2019/2022
Record Dates: First submitted 2021-02-14; First posted 2021-02-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Deficiency; Parkinson Disease
Keywords: parkinson's disease; deep brain stimulation; vitamin D; physical activity; functional tests; homocysteine; inflammatory markers; kynurenine pathway
MeSH Terms: conditions — Vitamin D Deficiency; Parkinson Disease; Motor Activity | interventions — Cholecalciferol; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The group will receive placebo treatment.
  Interventions: Drug: Placebo
- Vitamin D3 group (Experimental): The group will receive vitamin D3 supplementation.
  Interventions: Drug: Juvit D3

INTERVENTIONS:
Drug: Juvit D3 — Dosage based on the BMI as followed: for BMI under 25 - 4000 IU/day, for BMI between 25 and 30 - 5000 IU/day, and for BMI over 30 - 6000 IU/day.
  Other Names: vitamin D3
  Arms: Vitamin D3 group
Drug: Placebo — Matching amount of vegetable oil to the vitamin D3.
  Other Names: Vegetable oil
  Arms: Control group

SUMMARY:
Parkinson's disease (PD) is the second most frequently appearing neurodegenerative disease. It is a progressive disease of the central nervous system (CNS) and affects around 1% of people over 60 years old. During the progression decline of substantia nigra and deficits of dopamine are observed. The diagnosis is usually based on the motor symptoms such as resting tremor, bradykinesia, muscle stiffness, and postural instability. Common intercurrent symptoms are psychiatric problems like depression or dementia (1). Pharmacotherapy, for example, L-dopa or deep brain stimulation (DBS) are usually used to reduce the motor symptoms (2).

From many years the influence of insufficient vitamin D3 levels in human is investigated. In recent publications it was proved that the deficiency of vitamin D3 may lead to generation of reactive oxygen species that influence negatively on mitochondria. That may lead to increased muscle atrophy (3,4). Deficiency of vitamin D3 may be also connected with depression, dementia or the progression of neurodegenerative diseases (5). Moreover, recently studies proved that PD patients have low concentration of serum vitamin D3 (5), increased serum homocysteine (6) and abnormalities in kynurenine pathway (7).

It has beed proved that many forms of physical activity in PD patients improves mobility, static and dynamic balance but also may reduce the non-motor symptoms (8,9).

DETAILED DESCRIPTION:
Participants will be divided randomly into 2 groups: a control group and supplemented group.

Supplementation will last for 12 weeks.

Supplementation of vitamin D3 will be based on the participants Body Mass Index (BMI). The BMI will be measured by using the TANITA scale. The doses will be as followed: for BMI under 25 - 4000 International Units (IU)/day, for BMI between 25 and 30 - 5000 IU/day, and for BMI over 30 - 6000 IU/day. The placebo and control group will receive matching placebo treatment. Vitamin D3 as well as placebo will be in the same bottles with no labels on them.

Participants will be prompted to do 3500 steps per day in the first week of the research and finish the research with making 8000 per day. Participants will be obligated to measure the amount of steps by their phones.

There will be three meetings with the participants. On the first one there will be blood collection, participants will obtain questionnaires, about their daily activity and diet, to complete at home. Participants will have to sign the agreement of taking part in the research and perform functional tests. Also they will get their first supplementation bottles. On the second one the questionnaires will be collected, functional tests will be performed and supplementation will be replenished. On the third one the blood will be collected for the second time and functional tests will be performed again.

The questionnaire about daily activity will be International Physical Activity Questionnaire - Short Form.

The questionnaire about diet will be "Kwestionariusz QEB opracowany przez Zespół Behawioralnych Uwarunkowań Żywienia, Komitet Nauki o Żywieniu Człowieka, PAN". (Only polish version is available)

The blood will be collected into test tubes with clot activator, then centrifuged at 4000×g for 10 min at 4oC. The obtained serum samples will be stored in dark at -80oC until the analysis.

Investigators want to measure the changes in concentrations in blood of 25-hydroxycholecalciferol (25-OH D3), vitamin D3 binding protein, homocysteine, calcium, parathormone, interleukin-2 (IL-2), interleukin-6 (IL-6), interleukin-15 (IL-15), C-Reactive Protein (CRP), Tumor Necrosis Factor Alpha (TNF-α), serotonin, and the chosen markers of kynurenine pathway.

The functional tests will be assessed: 6 minute walk test (6MWT), test up&go (TUG) and 10 m walk test (10MWT). All tests will be performed in the on-phase of their usual anti-PD medications. All tests will be explained and demonstrated before they will be taken. If the first attempt will go well participant will follow to the next one. If any mistake will appear, participant will wait for a minute and try again. During every meeting the procedure of each test will be remind to the participants.

The 6MWT will be administered in a 15m line at the corridor. Participants will be instructed to go back and forth along without running the 15m line as far as they can in 6 min. The total distance will be measured after 6 min.

In TUG participants will be supposed to stand up from the chair, walk 3m, turn around, go back to the chair and sit down as fast as they can without running.

In 10MWT investigators will measure the time which takes the participants to walk through 10m form standing position.

ELIGIBILITY:
Inclusion Criteria:

* agreement to take part in a research,
* Subthalamic nucleus deep brain stimulation (STN-DBS) treatment,
* willingness to work.

Exclusion Criteria:

* supplementation of vitamin D before the research,
* serious comorbidity (like tumour, cerebrovascular disease, cardiorespiratory compromise, forced dementia).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The effects of vitamin D supplementation and physical activity on concentration of vitamin D3 in serum - the evaluation of changes before and after 12 weeks of supplementation and physical activity | The outcome measure will be assessed up to 1 year after the last participant will go under the second collection of blood.
  The blood will be collected two times - before the start of supplementation and physical activity and after 12 weeks of supplementation and physical activity - then the serum samples will be stored in -80oC before the analysis. Changes in concentration of vitamin D3 will be assessed by using liquid chromatography coupled with tandem mass spectrometry technique (LC-MS/MS).
The effects of vitamin D supplementation and physical activity on concentration of inflammatory markers in serum - the evaluation of changes before and after 12 weeks of supplementation and physical activity | The outcome measure will be assessed up to 1 year after the last participant will go under the second collection of blood.
  The blood will be collected two times - before the start of the supplementation and physical activity and after 12 weeks of supplementation and physical activity - then the serum samples will be stored in -80oC before the analysis. Changes in the concentration of IL-2, IL-6, IL-15, and TNF-α will be assessed by using a commercially available enzyme-linked immunosorbent assay (ELISA) kits.
The effects of vitamin D supplementation and physical activity on concentration of CRP in serum - the evaluation of changes before and after 12 weeks of supplementation and physical activity | The outcome measure will be assessed up to 1 year after the last participant will go under the second collection of blood.
  The blood will be collected two times - before the start of the supplementation and physical activity and after 12 weeks of supplementation and physical activity - then the serum samples will be stored in -80oC before the analysis. Changes in the concentration of CRP will be assessed by using a commercially available enzyme-linked immunosorbent assay (ELISA) kits.
The effects of vitamin D supplementation and physical activity on the 6 minute walk test - the evaluation of changes before and after 6 and 12 weeks of supplementation and physical activity | The outcome measure will be estimated up to 1 year after the last participant will perform the test on the last intervention.
  The test will be performed 3 time points. Before the supplementation and physical activity, after 6 week of supplementation and physical activity, and after 12 weeks of supplementation and physical activity. The distance covered by the participants will be measured each time and the analysis will be performed.
The effects of vitamin D supplementation and physical activity on the Test Up & Go and 10 meter walk test - the evaluation of changes before and after 6 weeks of supplementation and after 12 weeks of supplementation and physical activity | The outcome measure will be estimated up to 1 year after the last participant will perform the test on the last intervention.
  The Test Up & Go and 10 meter walk test will be performed 3 time points. Before the supplementation and physical activity, after 6 week of supplementation and physical activity, and after 12 weeks of supplementation and physical activity. The time achieved by the participants will be measured each time and the analysis will be performed.
The effects of vitamin D supplementation and physical activity on concentration of kynurenine pathway metabolites in serum - the evaluation of changes before and after 12 weeks of supplementation and physical activity | The outcome measure will be assessed up to 1 year after the last participant will go under the second collection of blood.
  The blood will be collected two times - before the start of supplementation and physical activity and after 12 weeks of supplementation and physical activity - then the serum samples will be stored in -80oC before the analysis. Changes in concentration of kynurenine pathway metabolites will be assessed by using liquid chromatography coupled with tandem mass spectrometry technique (LC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Zofia K Bytowska, MSc, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Background] da Silva AG, Leal VP, da Silva PR, Freitas FC, Linhares MN, Walz R, Malloy-Diniz LF, Diaz AP, Palha AP. Difficulties in activities of daily living are associated with stigma in patients with Parkinson's disease who are candidates for deep brain stimulation. Braz J Psychiatry. 2020 Apr;42(2):190-194. doi: 10.1590/1516-4446-2018-0333. Epub 2019 Aug 5. PMID 31389495
- [Background] Aum DJ, Tierney TS. Deep brain stimulation: foundations and future trends. Front Biosci (Landmark Ed). 2018 Jan 1;23(1):162-182. doi: 10.2741/4586. PMID 28930542
- [Background] Dzik KP, Kaczor JJ. Mechanisms of vitamin D on skeletal muscle function: oxidative stress, energy metabolism and anabolic state. Eur J Appl Physiol. 2019 Apr;119(4):825-839. doi: 10.1007/s00421-019-04104-x. Epub 2019 Mar 4. PMID 30830277
- [Background] Dzik KP, Skrobot W, Kaczor KB, Flis DJ, Karnia MJ, Libionka W, Antosiewicz J, Kloc W, Kaczor JJ. Vitamin D Deficiency Is Associated with Muscle Atrophy and Reduced Mitochondrial Function in Patients with Chronic Low Back Pain. Oxid Med Cell Longev. 2019 Jun 2;2019:6835341. doi: 10.1155/2019/6835341. eCollection 2019. PMID 31281588
- [Background] Pludowski P, Holick MF, Grant WB, Konstantynowicz J, Mascarenhas MR, Haq A, Povoroznyuk V, Balatska N, Barbosa AP, Karonova T, Rudenka E, Misiorowski W, Zakharova I, Rudenka A, Lukaszkiewicz J, Marcinowska-Suchowierska E, Laszcz N, Abramowicz P, Bhattoa HP, Wimalawansa SJ. Vitamin D supplementation guidelines. J Steroid Biochem Mol Biol. 2018 Jan;175:125-135. doi: 10.1016/j.jsbmb.2017.01.021. Epub 2017 Feb 12. PMID 28216084
- [Background] Licking N, Murchison C, Cholerton B, Zabetian CP, Hu SC, Montine TJ, Peterson-Hiller AL, Chung KA, Edwards K, Leverenz JB, Quinn JF. Homocysteine and cognitive function in Parkinson's disease. Parkinsonism Relat Disord. 2017 Nov;44:1-5. doi: 10.1016/j.parkreldis.2017.08.005. Epub 2017 Aug 9. PMID 28807493
- [Background] Sorgdrager FJH, Vermeiren Y, Van Faassen M, van der Ley C, Nollen EAA, Kema IP, De Deyn PP. Age- and disease-specific changes of the kynurenine pathway in Parkinson's and Alzheimer's disease. J Neurochem. 2019 Dec;151(5):656-668. doi: 10.1111/jnc.14843. Epub 2019 Aug 25. PMID 31376341
- [Background] Arfa-Fatollahkhani P, Safar Cherati A, Habibi SAH, Shahidi GA, Sohrabi A, Zamani B. Effects of treadmill training on the balance, functional capacity and quality of life in Parkinson's disease: A randomized clinical trial. J Complement Integr Med. 2019 Aug 21;17(1):/j/jcim.2019.17.issue-1/jcim-2018-0245/jcim-2018-0245.xml. doi: 10.1515/jcim-2018-0245. PMID 31433785
- [Background] Brienesse LA, Emerson MN. Effects of resistance training for people with Parkinson's disease: a systematic review. J Am Med Dir Assoc. 2013 Apr;14(4):236-41. doi: 10.1016/j.jamda.2012.11.012. Epub 2013 Jan 11. PMID 23318666